CLINICAL TRIAL: NCT01285375
Title: Safety and Preliminary Efficacy of the Treatment of Kidney Allografts With Curcumin-containing Preservation Solution
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Academy of Finland (Other)
Responsible Party: Kaija Salmela, MD, Head of Kidney Transplantation Unit, Department of Liver and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 236153; 236153 (Registry Identifier: Hospital District of Helsinki and Uusimaa)
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: End Stage Renal Failure With Renal Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDC graft perfusion (Active Comparator): Flushing of kidney allografts prior to transplantation with UW-solution containing CDC
  Interventions: Device: CDC solution
- Sham perfusion (Sham Comparator)
  Interventions: Device: UW-solution

INTERVENTIONS:
Device: CDC solution — 2 ml of CDC 12/mg/ml is added to 1 l of UW solution. 500 ml of of this solution is used for flushing the kidney allograft prior to transplantation
  Other Names: Curcumin-cyclodextrin
  Arms: CDC graft perfusion
Device: UW-solution — 500 ml of UW solution is used for flushing the kidney allograft prior to transplantation
  Other Names: Viaspan
  Arms: Sham perfusion

SUMMARY:
The safety and preliminary efficacy of the addition of an aqueous curcumin-cyclodextrin complex (CDC) solution to graft perfusion solution is studied. CDC has proved safe and highly effective in preventing primary graft non-function, delayed graft function and chronic dysfunction in pre-clinical kidney transplantation animal models. The hypothesis is that addition of CDC to the graft perfusion solution will decrease the incidence of delayed graft function in human kidney transplantation subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD assigned for kidney transplantation, written informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Delayed Graft Function | 7 days

SECONDARY OUTCOMES:
Primary non-function | 1 year
Acute rejection | 1 year
Graft function eGFR | 30 days, 90 days
Graft Survival | 1 year
Patient Survival | 1 year
Length of stay in hospital | upto 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kaija Salmela, Docent, Principal Investigator — Head of Kidney Transplantation Unit
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland